CLINICAL TRIAL: NCT02134405
Title: Rebamipide in Combination With Esomeprazole in the Management of Asian Patients With Functional Dyspepsia: a Multi-national, Randomised, Double-blind, Placebo-controlled Study
Brief Title: Rebamipide in Combination With Esomeprazole in the Management of Asian Patients With Functional Dyspepsia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Collaborators: Zhejiang Provincial Hospital of TCM (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 037-OTC-1203i
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Dyspepsia
Keywords: functional dyspepsia; symptoms; proton pump inhibitor; gastritis
MeSH Terms: conditions — Dyspepsia; Gastritis | interventions — rebamipide; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rebamipide and Esomeprazole (Experimental): Rebamipide tablets 100mg tid for 8 weeks Esomeprazole tablets 20mg od for 8 weeks
  Interventions: Drug: Rebamipide; Drug: Esomeprazole
- Rebamipide and placebo (Active Comparator): Placebo drug with Rebamipide 100mg tid
  Interventions: Drug: Rebamipide; Drug: Placebo (for Esomeprazole)

INTERVENTIONS:
Drug: Rebamipide — Rebamipide 100mg tid
  Other Names: Mucosta
Drug: Placebo (for Esomeprazole) — Sugar pill manufactured to mimic Esomeprazole
  Other Names: placebo
  Arms: Rebamipide and placebo
Drug: Esomeprazole — Esomeprazole tablets 20mg o.d. for 8 weeks
  Other Names: Nexium
  Arms: Rebamipide and Esomeprazole

SUMMARY:
This is a multi-Asian-centre randomised controlled trial of Rebamipide alone vs Rebamipide with Esomeprazole in the treatment of adult patients with Functional Dyspepsia. The hypothesis is that a combination therapy is superior to mono-therapy in the control of patients' symptoms and quality of life improvement.

DETAILED DESCRIPTION:
Primary Objective: To assess the efficacy of Rebamipide in combination with Esomeprazole in the improvement of symptoms of Functional Dyspepsia in Asian patients compared to Esomeprazole alone Secondary Objective: i. To assess the efficacy of Rebamipide in combination with Esomeprazole in the improvement of quality of life in Asian patients with Functional Dyspepsia compared to Esomeprazole alone ii. To assess the cost-effectiveness of Rebamipide in combination with Esomeprazole compared to Esomeprazole alone after 8, 12 weeks of treatment iii. To assess the safety of Rebamipide in combination with Esomeprazole in adults with functional dyspepsia after 8 weeks of treatment.

Trial Design Multi-national, randomised, double-blind, placebo-controlled study

Treatment Group:

* Study Group: Rebamipide + Esomeprazole
* Control Group: Rebamipide placebo + Esomeprazole Investigational Product (IP): Rebamipide 100 mg tablet Rebamipide placebo tablet Esomeprazole 20 mg tablet Dosage regimen: Administration route: PO Rebamipide 100 mg t.i.d Rebamipide placebo t.i.d Esomeprazole 20 mg o.d Target Population Male or female subjects aged from 18 years to less than 80 years with a diagnosed of Functional Dyspepsia (FD) Primary Endpoint: Change in Leeds Dyspepsia Questionnaire (LDQ) total score from baseline to 8 weeks of treatment Secondary Endpoints: 1. The change in Health-Related Quality of Life (EQ-5D) from baseline to 8 weeks of treatment 2. The cost effectiveness based on cost per QALY gained between the study group compared to the control group at 8, 12 weeks 3. The change in Leeds Dyspepsia Questionnaire (LDQ) total score and Health-Related Quality of Life (EQ-5D) from baseline to 12 weeks Inclusion Criteria: 1. Patients diagnosed with Functional Dyspepsia using Rome III diagnostic criteria 2. Age ≥ 18 years, < 80 years 3. Subject who has ability to provide written informed consent and willingness to comply with the requirement of the protocol 4. Able to communicate in English, Malay or Mandarin languages 5. Patients on prior dyspepsia treatment - after washout period of 1 week Exclusion Criteria: 1. Patients with known hypersensitivity to Rebamipide and/or Esomeprazole and any other component of these formulations.

  2. Pregnant, nursing, and childbearing potential women who is unwilling to effective contraception; for example, oral contraceptives, hormonal methods, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods (i.e., condom or occlusive cap with spermicidal foam/gel/film/cream/ suppository), male sterilization, and true abstinence 3. Presence of family history of GI malignancy or alarm features suggested malignancy - e.g. Unintentional weight loss (more than 10% of body weight in recent 6 months), GI bleeding 4. Patients consuming regular Aspirin or NSAIDs (except low-dose Aspirin at a dose of 325 mg/day or less for cardiovascular prophylaxis) 5. History of erosive esophagitis, peptic ulcer disease within 1 year prior to the screening 6. History of gastrointestinal (GI) malignancy, primary esophageal motility disorder, documented upper GI surgery 7. Patients with any hepatobiliary or pancreatic diseases 8. Patients with severe depression, anxiety, or other psychological disorder 9. Patients with any terminal disease 10. Presence of irritable bowel syndrome (Rome III criteria) or inflammatory bowel disease (IBD) 11. Necessary to have a continuous concomitant treatment with sucralfate, quinidine, warfarin, phenytoin, bisphosphonates, methotrexate, ketoconazole, fluconazole, itaconazole, diazepam, anti-cholinergics, H2RAs, PPIs (except study drug), prokinetics, and/or NSAIDs (except topical use of NSAIDs; in systemic NSAIDs ≤2 days/week) 12. Use of PPIs (except study drug), H2RAs, prokinetics, antibiotics (except topical use), misoprostol, or bismuth compounds within 1 week prior to the screening, and who were taking antibiotics used to eradicate Helicobacter pylori within 4 weeks prior to the screening 13. Unable to communicate in English, Malay, or Mandarin 14. Other conditions determined by the investigator to be inappropriate for this clinical study Duration of treatment: 8 weeks Number of subjects: Ninety-three patients per each group with 90% power at the 0.05 significance level were used. Considering 10% drop-out rate, total of 208 patients (104 patients per each group) will be enrolled in the study.

Total: 208 Study Group: 104 Control Group: 104 Anticipated Timelines: Duration of trial: 18 months Start of recruitment: March 2014 End of recruitment: August 2015 Last subject out: Oct 2015

Statistical Methodology:

Primary Endpoint Change in Leeds Dyspepsia Questionnaire (LDQ) total score from baseline to 8 weeks of treatment

Secondary Endpoint

1. The change in Health-Related Quality of Life (EQ-5D) from baseline to 8 weeks of treatment
2. The cost effectiveness based on cost per QALY gained between the study groups compared to the control group at 8, 12 weeks
3. The change in Leeds Dyspepsia Questionnaire (LDQ) total score and Health-Related Quality of Life (EQ-5D) from baseline to 12 weeks

Summary statistics of the endpoints will be provided. Mean change will be evaluated by two sample t-test or Wilcoxon's rank sum test according to the normal distribution of analyzed variable.

Safety Endpoint

1. Adverse events The number of cases of AEs and the proportion of patients who experienced AEs will be summarized by descriptive statistics (frequency and proportion) for each study group.
2. Laboratory Test and Vital Signs All laboratory values and vital signs will be compared within study group and between study groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Functional Dyspepsia using Rome III diagnostic criteria
2. Age ≥ 18 years, < 80 years
3. Subject who has ability to provide written informed consent and willingness to comply with the requirement of the protocol
4. Able to communicate in English, Malay or Mandarin languages
5. Patients on prior dyspepsia treatment - after washout period of 1 week

Exclusion Criteria:

1. Patients with known hypersensitivity to Rebamipide and/or Esomeprazole and any other component of these formulations.
2. Pregnant, nursing, and childbearing potential women who is unwilling to effective contraception; for example, oral contraceptives, hormonal methods, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods (i.e., condom or occlusive cap with spermicidal foam/gel/film/cream/suppository), male sterilization, and true abstinence
3. Presence of family history of GI malignancy or alarm features suggested malignancy - e.g. Unintentional weight loss (≥ 10% of body weight in recent 6 months), GI bleeding
4. Patients consuming regular Aspirin or NSAIDs (except low-dose Aspirin at a dose of 325 mg/day or less for cardiovascular prophylaxis)
5. History of erosive esophagitis, peptic ulcer disease within 1 year prior to the screening
6. History of gastrointestinal (GI) malignancy, primary esophageal motility disorder, documented upper GI surgery
7. Patients with any hepatobiliary or pancreatic diseases
8. Patients with severe depression, anxiety, or other psychological disorder
9. Patients with any terminal disease
10. Presence of irritable bowel syndrome (Rome III criteria) or inflammatory bowel disease (IBD)
11. Necessary to have a continuous concomitant treatment with sucralfate, quinidine, warfarin, phenytoin, bisphosphonates, methotrexate, ketoconazole, fluconazole, itaconazole, diazepam, anti-cholinergics, H2RAs, PPIs (except study drug), prokinetics, and/or NSAIDs (except topical use of NSAIDs; in systemic NSAIDs ≤2 days/week)
12. Use of PPIs (except study drug), H2RAs, prokinetics, antibiotics (except topical use), misoprostol, or bismuth compounds within 1 week prior to the screening, and who were taking antibiotics used to eradicate Helicobacter pylori within 4 weeks prior to the screening
13. Unable to communicate in English, Malay, or Mandarin
14. Other conditions determined by the investigator to be inappropriate for this clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Dyspepsia symptoms | 8 weeks
  To assess the efficacy of Rebamipide in combination with Esomeprazole in the improvement of symptoms of Functional Dyspepsia in Asian patients compared to Esomeprazole alone.

SECONDARY OUTCOMES:
quality of life | 8 weeks
  i. To assess the efficacy of Rebamipide in combination with Esomeprazole in the improvement of quality of life in Asian patients with Functional Dyspepsia compared to Esomeprazole alone

OTHER OUTCOMES:
Financial costs | 12 weeks
  To assess the cost-effectiveness of Rebamipide in combination with Esomeprazole compared to Esomeprazole alone after 8, 12 weeks of treatment
Adverse events | 12 weeks
  To assess the safety of Rebamipide in combination with Esomeprazole in adults with functional dyspepsia after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Mahadeva, MRCP, MD, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia